CLINICAL TRIAL: NCT06659796
Title: LifeVac Survey Study
Status: Completed | Type: Observational
Sponsor: LifeVac, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-001
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Airway Obstruction; Choking
Keywords: Airway obstruction; Choking
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Users of LifeVac device: Individuals who have used the LifeVac device during a choking emergency
  Interventions: Device: LifeVac

INTERVENTIONS:
Device: LifeVac — Removal of airway obstruction during choking emergency

SUMMARY:
This observational, non-interventional survey study is intended to explore user experiences with the LifeVac airway clearance device, with a particular emphasis on real-world application in choking emergencies in the USA. This study seeks to gather valuable insights from a representative sample of the LifeVac device purchaser base.

The main questions the study aims to answer are:

1. Is the LifeVac device safe for individuals experiencing a choking emergency?
2. Is the LifeVac device successful in removing an obstruction during a choking incident?

Participants: Purchasers of the LifeVac device.

DETAILED DESCRIPTION:
Foreign Body Airway Obstruction (FBAO), commonly referred to as choking, occurs when an aspirated solid or semisolid object becomes lodged in a person's larynx or trachea. If the object is large enough it may cause the complete (or near complete) obstruction of the airway. Without oxygen, brain damage can occur in as soon as four minutes following the event.

LifeVac is a non-powered, non-invasive, single-use airway clearance device developed for resuscitating a victim with an airway obstruction when current choking protocols (basic life support [BLS]) failed to remove the obstruction. The device is intended be used on adults and children, in home and non-home settings, and can be administered by professional/HCP users or laypersons without professional training in a choking emergency.

This observational, non-interventional survey study will be conducted on purchasers of the LifeVac device. The study intends to obtain responses from at least 26 users of the device in each of the two age groups of interest, individuals up to 19 years of age (pediatric) and above 20 years of age (adult), and capture unbiased information on the device users' experience, regardless of its outcome.

Objectives:

1. Gather information on device usage patterns and user experiences with the LifeVac airway clearance device.
2. Collect data on the safety and effectiveness of the device in real-world choking interventions.

Target Population:

Purchasers of the LifeVac device in the USA from 2015 to April 2024.

Data Collection Procedure:

1. Purchasers will be invited to participate via a standardized email with a link to an online platform (IntelliSurvey, Inc.) independent of the device manufacturer.
2. Participation will require electronic consent before accessing the survey.
3. The survey is accessible through a web browser and can be completed on a desktop computer or mobile device.

ELIGIBILITY:
Inclusion Criteria:

* Purchases of the LifeVac device Original database: all purchasers of the LifeVac device from the LifeVac website starting in 2015 until April 2024, a timeframe that yields a database of above 450,000 individuals with no email duplications and third party suppliers.

Survey batches: randomly selected sample of 50,000 purchasers (10% of the database).

Number of batches required will be based on response rate.

* English speaking
* Ability to understand and accept the consent form

Exclusion Criteria:

* Did not purchase a LifeVac device
* Third party suppliers
* Non-English speakers (as LifeVac labeling and survey materials are only available in English)
* Unwilling or unable to accept the consent form

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • Purchasers of the LifeVac device in the USA from 2015 to April 2024
Sampling Method: Probability Sample
Enrollment: 2930 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Up to 1 week
  Occurrence of any serious adverse events (SAE) associated with the use of the LifeVac device.
Primary Effectiveness Endpoint | Up to 1 week
  Confirm success or partial success in relieving airway obstruction in at least 80% of uses of the device.

SECONDARY OUTCOMES:
Secondary Safety Endpoint | Up to 1 week
  Occurrence of any adverse events (AE) associated with the use of the LifeVac device.
Secondary Effectiveness Endpoint | Up to 1 week
  Explore potential correlations between the outcome of the device use with age of the choking person, the nature of the obstruction, and the environment where the choking incident transpired.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Nadai, Principal Investigator — Boston MedTech Advisors
Locations (1):
- Boston MedTech Advisors, Dedham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No